CLINICAL TRIAL: NCT05935020
Title: Feasibility of a Randomized Trial Comparing Exercise-based Rehabilitation With Non-exercise-based Recovery After Total Knee Arthroplasty; DRAW-TKA Hybrid 1 Feasibility Trial
Brief Title: Does Rehabilitation After Total Knee Arthroplasty Work? - Feasibility Trial
Acronym: DRAW-TKA-Fea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Collaborators: Danske Fysioterapeuter (Other); Sygekassernes Helsefond (Other); University of Copenhagen (Other); The Danish Rheumatism Association (Other); Tværspuljen (Unknown)
Responsible Party: Principal Investigator, Birk Mygind Grønfeldt, PhD Fellow, Copenhagen University Hospital, Hvidovre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: DRAW-TKA-Feasibility
Record Dates: First submitted 2023-06-26; First posted 2023-07-07 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-02

CONDITIONS: Osteoarthritis, Knee
Keywords: Total Knee Replacement; Osteoarthritis, Knee; Exercise-based Rehabilitation
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Two group, parallel, randomized, controlled feasibility trial
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigator and Outcomes Assessor are blinded to participant group allocation. Further, the personnel administering the intervention after discharge from the surgical ward (Care Provider) is masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (Active Comparator): Referral to municipal rehabilitation after TKA
  Interventions: Other: Usual care - Municipal exercise-based rehabilitation; Behavioral: Symptom guide and encouragement to follow DHA/WHO recommendations for physical activity
- Return to Everyday Life (Other): No referral to municipal rehabilitation after TKA
  Interventions: Other: Return to Everyday life; Behavioral: Symptom guide and encouragement to follow DHA/WHO recommendations for physical activity

INTERVENTIONS:
Other: Usual care - Municipal exercise-based rehabilitation — The patients in this group follow prescribed (by the orthopedic surgeon) "usual care" municipal exercise-based rehabilitation. The content of the rehabilitation is planned in collaboration between the patient and the physical therapist, based on the offered municipal treatment options (which varies between municipalities) and patient preferences (i.e., home-based exercise, outpatient exercise, group-based exercise, or a combination thereof). The contents of the municipal services offered will be described in detail in the trial report.
  A prescribed therapeutic rehabilitation exercise plan could for instance be a 6-week combined home-exercise (1-2 times/week) and group-exercise (1 time/week) intervention, followed by encouragement to continue self-administered home exercise after the 6 weeks.
  Other Names: Referral to Municipal Rehabilitation after Surgery
  Arms: Usual Care
Other: Return to Everyday life — The patients in this group return to their desired pre-surgical activities, at their own speed, when they feel that they are ready for it. They are not prescribed any exercise-based rehabilitation (usual care) by their orthopedic surgeon.
  This effectively means they will not receive a therapeutic progressive exercise plan; designed and prescribed to restore previous function or reducing pain or disability caused by injury, disease, or surgery - typically referred to as "exercise therapy" or "therapeutic exercise".
  Other Names: No referral to municipal rehabilitation after surgery
  Arms: Return to Everyday Life
Behavioral: Symptom guide and encouragement to follow DHA/WHO recommendations for physical activity — Participants in both groups receive a recovery-guide pamphlet at discharge, containing the following information: 1) Recommendations to follow DHA/WHO guidelines for physical activity, 2) Figures and tables describing common post-operative symptoms (symptom guide), and when to react (when the symptoms may require attention from a health-professional), 3) What to expect from the post-surgical period in relation to activities of daily living, 4) Common short- and long-term complications to total knee arthroplasty and 5) Trial-participant and ethics-committee information documents. Parts 2-4 are usual clinical practice, with slight variations in descriptions between sites.
  After surgery, participants in both groups are encouraged to resume their desired pre-surgical activities when they feel they are able (within the limits given from the orthopedic wards).
  Other Names: Symptom self-management and encouraged physical activity

SUMMARY:
The aim of this feasibility trial is to investigate the feasibility of a trial intervention for a population of patients after total knee replacement for osteoarthritis. This study follows a hybrid type 1 design where the primary focus is on the feasibility of the intervention, and the secondary focus is on gaining a better understanding of context and acceptability.

The main questions it aims to answer are:

* Recruitment (Process/Resources): Are patients willing to engage, and stay, in the trial (estimated by inclusion-rate, participant retention, etc.) and what reasons do patients give for not wishing to enroll or later dropping out of the trial? (inquired face-to-face, during enrolment).
* Harms (Scientific): Does the non-exercise intervention appear "safe" (i.e. not harmful) for the patients? (estimated by for instance: adverse events, reasons for dropouts and sense of security).
* Trial procedure feasibility (Management/Scientific): How well does recruitment and trial procedures work at trial sites? (estimated through feedback from site personnel).
* Participant (patient) experienced acceptability of their assigned intervention: An interview-based follow-up using the Theoretical Framework of Acceptability.

Participants will be randomized to one of two interventions, at discharge from the hospital, following knee replacement, which are being tested for feasibility:

1. "Usual-care" - referral to municipal (free-of-charge) physiotherapy (commonly 6-8 weeks of therapeutic exercise).
2. "Return to everyday life" - no referral to municipal physiotherapy.

Participants in both groups are encouraged to follow WHO guidelines of physical activity, to the degree that their post-surgical symptoms allow (within their orthopedic surgeon's recommendations/limitations). All participants are given a "symptom guide", meaning a folder containing information on what to expect, and when and what to react to, during their recovery after the knee-replacement.

For clarity it should be mentioned, that the quantitative and qualitative data-outputs will be reported separately for improved clarity (the study is not a mixed methods design).

DETAILED DESCRIPTION:
Feasibility-criteria (Handling of feasibility outcomes: primary and secondary):

As the feasibility-trial investigates a combination of randomization acceptance, trial procedures, and intervention organization, a primary outcome measure is not specified. The outcome measures planned in the large scale effectiveness trial will be applied, but the outcomes will not be used to assess efficacy, as the trial is not powered for these outcomes. They will be used to indicate efficiency of trial procedures and safety, and to gain information on patients' willingness to enroll and remain in the trial.

Feasibility outcomes will be assessed when all 24 feasibility participants have completed their 12-week follow-up outcome-assessment. An overall assessment of large-scale trial feasibility will be made in the main investigator group, by comparing feasibility research questions with feasibility criteria/outcomes. As there are many components within the feasibility criteria, a summary of findings will be produced. This is used to inform a discussion (main investigator group) to find consensus regarding a final decision on whether a large-scale trial is considered feasible (see Criterion interpretation below).

The feasibility components are organized as related to process, resources, management and scientific, as proposed by Thabane (Thabane et al., 2010). The recruitment (process and resources) is considered the primary feasibility outcome and thusly has specified feasibility criteria.

Criterion interpretation:

It should be noted that feasibility criteria are set to inform a basis for discussion of the trial feasibility in the main investigator group, and the final interpretation is based on the discussion (mentioned above) of which criteria succeeded, which failed, and to which degree. Thusly, a single criterion exactly exceeding or staying just below the criteria set is still subject to discussion and may not singularly mean that the large-scale trial is not feasible (i.e., having only 84% of participants complete the primary outcome does not automatically cancel the large-scale trial, nor does a 85% primary outcome completion rate make the criteria exempt from a discussion regarding feasibility). The trial group discussion aims to result in one of the following interpretations (with elaboration where needed):

1) main study not feasible - stop main study, 2) feasible with modification - continue main study with modifications, 3) feasible without modification - no modifications but close monitoring, 4) feasible as is - continue without modifications.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Residing in one of fourteen collaboration municipalities
* Referral to primary total knee arthroplasty for osteoarthritis

Exclusion Criteria:

* Insufficient danish skills (read/write/speak) to understand questionnaires and outcomes
* Inability to provide informed consent
* Severe surgical sequelae (i.e. requiring revision surgery, joint mobilization under anaestesia, or joint infection)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-08-22 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Feasibility Trial - Primary outcome is an evaluation of trial feasibility: | Full duration of feasibility trial from enrollment to last follow-up at 12 weeks from surgery
  The following criteria are considered most important to evaluate feasibility:
  * No more than 20% of participants may drop out of the "return-to-everyday-life" group because they change their mind and wish to receive exercise-based rehabilitation instead (wish to cross over)
  * At least 10% of the patients who receive full trial information, are subsequently enrolled in the trial
  * At least 85% of enrolled participants complete the primary outcome assessment at 12 weeks
  * At least one participant (on average) must be included at each site, each week
  The criteria, and and all other outcomes, form the basis of a trial group discussion with the intent of agreeing on one of the following interpretations (large-scale trial feasibility):
  1) Main study not feasible - stop main study, 2) Feasible with modification - continue main study with modifications, 3) Feasible without modification - no modifications but close monitoring, 4) Feasible as is - continue without modifications.
Recruitment (Process and resources): | Full duration of feasibility trial from enrollment to last follow-up at 12 weeks from surgery
  * Enrolment rate - how many of the eligible patients (given full trial information) end up as participants (signed informed consent)
  * Barriers to participation - why do patients decline to enroll (enquired when they decline participation when given full trial information)
  * Retention rate - how many participants complete the 12-week follow-up
  * Barriers to retention - why do participants decide to discontinue participation in the trial
  * Eligibility criteria - how many participants drop out after enrolment
  * Trial measures - how many participants have blank/incomplete/complete tests and questionnaires

SECONDARY OUTCOMES:
Harms (Scientific) | Full duration of feasibility trial from enrollment to last follow-up at 12 weeks from surgery
  Number and reasons for dropouts and/or adverse events will be closely monitored during the feasibility-trial, to ensure that patients are not subjected to a potentially harmful intervention (or non-intervention).
  Though the feasibility trial is underpowered (too few participants) to be conclusive regarding harms/safety, this will be monitored to indicate risks.
  If the within-group response at follow-up (12 weeks) indicates a negative effect of at least the minimal clinically important difference on outcomes (i.e. more pain and/or worsening of symptoms) compared to baseline, without other explanatory factors (i.e. infection or other surgical sequelae), the safety and ethics of continuing of the intervention in the effect trial will be evaluated in the trial team.
Trial personnel feasibility (Management/Scientific) | Full duration of feasibility trial from enrollment to last follow-up at 12 weeks from surgery
  The trial personnel feasibility is assessed by scheduled, informal interviews with trial personnel, to uncover potential problems and to have feedback on trial procedures. Questions for these interviews are based on the following suggested questions for type 1 hybrid designs (Curran et al., 2012):
  * What are potential barriers and facilitators to "real-world" implementation of the intervention?
  * What problems were associated with delivering the intervention during the clinical effectiveness trial and how might they translate or not to real-world implementation?
  * What potential adaptations to the clinical intervention could be made to maximize implementation?
  * What potential implementation strategies appear promising?
  This will relate to how the personnel experience the trial procedures being an obstruction during clinical routine tasks and/or obstacles that can impact the methodological quality.
Participant symptom guide follow-up | Full duration of feasibility trial from enrollment to last follow-up at 12 weeks from surgery
  As the symptom guide is intended to assist participants with symptom guidance, it is important to assess whether the participants have used it (received it) and how. Therefore, all participants will be enquired whether they received the symptom-guide and other trial materials, how they used it and what they like/dislike about it.
Participant (patient) experiences and experienced acceptability; of their allocated intervention | Interviews will be conducted after participants complete the 12 week follow-up
  Following completion of the 12 week follow-up, participants are encouraged to engage in interviews to assess their experiences and their experienced acceptability of the trial intervention they were randomly allocated. The interview guide is built on the Theoretical Framework of Acceptability of interventions (TFA), an is planned analysed using the same framework.
  The acceptability interviews may provide relevant patient perspectives on trial procedures, participant documents etc. These acceptability findings are considered relevant outcomes to the feasibility trial (and a possible following large scale effectiveness trial), although planned reported in separate papers.
  This outcome will be reported on separately from the remaining feasibility outcomes, to more concisely describe methods used for each type of data (qualitative or quantitative).

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Copenhagen University Hospital Hvidovre, Hvidovre
  - Næstved Sygehus, Næstved

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD.

REFERENCES:
- [Derived] Gronfeldt BM, Skou ST, Kirk JW, Troelsen A, Bandholm T; DRAW-TKA collaborator group. Feasibility of a randomized trial comparing exercise-based rehabilitation to no exercise-based rehabilitation after total knee arthroplasty: DRAW-TKA hybrid 1 RCT. Osteoarthr Cartil Open. 2025 Nov 21;8(1):100708. doi: 10.1016/j.ocarto.2025.100708. eCollection 2026 Mar. PMID 41431738